CLINICAL TRIAL: NCT03408145
Title: Short-Term Changes in Knee Synovial Fluid Composition Following Intraarticular Implantation of Amniotic Tissue Allograft
Brief Title: Stem Cell and Growth Factor Injury and Arthritis Clinical Research Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Stone Research Foundation for Sports Medicine and Arthritis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: SRF-037
Record Dates: First submitted 2018-01-08; First posted 2018-01-23 (Actual); Last update posted 2021-03-25 (Actual); Status verified 2020-06

CONDITIONS: Osteoarthritis, Knee
Keywords: Stem Cell Therapy; Injection; Hyaluronic Acid; Synovial Fluid
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Viscosupplementation; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Saline (Placebo Comparator): The investigators aspirate 1-2ml of Synovial Fluid from the knee joint prior to administering a series of four injections (2.5ml, 2.5ml, 2.5ml and 1ml of Saline) comprising a total volume of 8.5ml fluid during one procedure.
  Interventions: Drug: Saline
- Hyaluronic Acid & Saline (Active Comparator): The investigators aspirate 1-2ml of Synovial Fluid from the knee joint prior to administering a series of four injections (2.5ml, 2.5ml, 2.5ml of Hyaluronic Acid and 1ml Saline) comprising a total of 8.5mL fluid during one procedure.
  Interventions: Device: Hyaluronic Acid; Drug: Saline
- Amniotic Tissue & Saline (Active Comparator): The investigators aspirate 1-2ml of Synovial Fluid from the knee joint prior to administering a series of four injections (2.5ml, 2.5ml, 2.5ml of Saline and 1ml Amniotic Tissue Allograft) comprising a total of 8.5mL fluid during one procedure.
  Interventions: Device: Amniotic Tissue Allograft
- Amniotic Tissue & Hyaluronic Acid (Experimental): The investigators aspirate 1-2ml of Synovial Fluid from the knee joint prior to administering a series of four injections (2.5ml, 2.5ml, 2.5ml of Hyaluronic Acid and 1ml Amniotic Tissue Allograft) comprising a total of 8.5mL fluid during one procedure.
  Interventions: Device: Hyaluronic Acid; Device: Amniotic Tissue Allograft

INTERVENTIONS:
Device: Hyaluronic Acid — Injection of 3x 2.5ml of Hyaluronic Acid
  Other Names: Viscosupplementation; Supartz
  Arms: Amniotic Tissue & Hyaluronic Acid; Hyaluronic Acid & Saline
Device: Amniotic Tissue Allograft — Injection of 1x 1ml of Amniotic Tissue Allograft
  Other Names: Stem Cells; Growth Factors; Palingen InovoFLo
  Arms: Amniotic Tissue & Hyaluronic Acid; Amniotic Tissue & Saline
Drug: Saline — Injection of Saline
  Other Names: Sodium Chloride; NaCl
  Arms: Hyaluronic Acid & Saline; Saline

SUMMARY:
The investigators believe that amniotic tissue allografts may be an effective modality to treat osteoarthritis (OA) of the knee. One important mechanism of action may be stimulation of the synovial cells to increase production of endogenous hyaluronic acid (HA). A second mechanism may be the increase in the anabolic factors and a decrease in degenerative factors in the joint. The Investigators propose to quantify the concentration of HA and selected anabolic and degradative factors in synovial fluid aspirate pre and post implantation. While the treatment provided is designed to provide pain relief for symptoms, the purpose of this study is to learn more information about the impact of amniotic tissue allografts on inflammatory markers and growth factors in the knee joint.

DETAILED DESCRIPTION:
The investigators believe that amniotic tissue allografts may be an effective modality to treat osteoarthritis (OA) of the knee. One important mechanism of action may be stimulation of the synovial cells to increase production of endogenous hyaluronic acid (HA). A second mechanism may be the increase in the anabolic factors and a decrease in degenerative factors in the joint. The Investigators propose to quantify the concentration of HA and selected anabolic and degradative factors in synovial fluid aspirate pre and post implantation. While the treatment provided is designed to provide pain relief for symptoms, the purpose of this study is to learn more information about the impact of amniotic tissue allografts on inflammatory markers and growth factors in the knee joint.

The purpose of this study is to determine the changes in the composition of synovial fluid resulting from implantation of amniotic tissue allograft in the knee.

This study will characterize the chemical profile of painful osteoarthritic joints and the influence of various injections containing cells and/or growth factors on that chemical profile. The addition of amniotic tissue allograft to HA injections may be an, effective treatment for people with knee pain resulting from OA and furthermore may lead to customization and/or the identification of the most efficacious combination of joint injections.

Prior to any study-related treatment, participants will undergo an Institutional Review Board (IRB)-approved informed consent process for aspiration of synovial fluid, followed by a randomized injection of either A) saline only, B) hyaluronic acid, C) amnionic allograft, or D) hyaluronic acid plus amnionic allograft, with a second aspiration performed 1 week after injection. Synovial fluid samples from 88 participants indicated for amniotic tissue implantation will be analyzed in vitro to determine the cellular and biochemical characterization of the fluid obtained.

The aim of this study is to determine the changes in composition of synovial fluid resulting from implantation of amniotic tissue allograft in the knee. There is always a possibility that the insertion of a needle may in itself result in a change in the composition of synovial fluid and therefore to increase the strength of the study control arm (placebo) is necessary. The placebo controlled group is justified to provide evidence that the standard of care and research treatments are safe and efficacious.

Participants will be randomly assigned to one of four treatment groups:

Group A: Placebo - saline Group B: Standard of care treatment - hyaluronic acid, Group C: Standard of care treatment - amnionic allograft, or Group D: Research treatment: hyaluronic acid plus amnionic allograft.

Prior to undergoing treatment, participants will be asked to complete a series of subjective health questionnaires. Upon completion of the questionnaires, a 1-2mL sample of synovial fluid will be aspirated from each subject. The collection of the synovial fluid is performed strictly for research purposes related to this study. Treatment will be administered according to the group the participant was randomly assigned to.

One week (+/- 3 days) following the treatment, the participant will return to the clinic, and will complete a second set of questionnaires, after which a second aspiration of 1-2mL of synovial fluid will be taken. If the participant received a placebo injection (saline only), they will be given an opportunity to receive an amniotic tissue allograft injection and/or hyaluronic acid .

Participation in this study will require that the investigators perform some procedures in addition to the standard of care. Standard of care is defined as:

* Receipt of a therapeutic injection of hyaluronic acid or implantation of amniotic tissue allograft
* Completion of subjective outcome questionnaires prior to treatment

Research specific procedures are defined as:

* Aspiration of knee synovial fluid during treatment
* Aspiration of knee synovial fluid one week after treatment
* Completion of subjective outcome questionnaires at one week following treatment
* Analysis of knee synovial fluid for increased levels of anabolic factors, IL1ra, TMP1, TMP2, HA, and IGF1 as well as decreased levels of degradative factors, IL-1, TNF-alpha, IL-10, MMP-2, MMP-9, TGF-beta

ELIGIBILITY:
Inclusion Criteria:

1. Patients age 18 and over
2. Previous diagnosis of knee OA,
3. Kellgren-Lawrence grade of 2 - 4
4. Minimum Visual Analogue Scale (VAS) pain score of 3 on a scale of 0 - 10 where 0 is no pain and 10 is the highest level of pain
5. Can give written informed consent

Exclusion Criteria:

1. Receipt of HA, Platelet Rich Plasma (PRP) or amniotic cell injections in the previous 6 months
2. Recent history of surgery to the same joint in the previous 3 months
3. A clinical diagnosis of inflammatory arthritis made by history, examination or serology
4. An active or latent infection of the affected knee joint or any other systemic infection currently under treatment or treated within the previous 3 months
5. A history of chronic alcohol or drug abuse during the six months prior to the study
6. Clinically documented acute or unstable concomitant disease, other than the condition to be treated in this study that might be a confounding reason for the presence of pathogens (i.e. renal, hepatic, cardiac, endocrine, hematologic, autoimmune, metabolic bone, crystal deposition, severe degenerative joint, neoplastic diseases)
7. Systemic or intra-articular administration, within twenty days prior to the procedure, of any type of corticosteroids, antineoplastic, immune stimulating or immunosuppressive agents
8. Participation in any other investigational drug or device trial during the 30 days prior to screening visit or who will receive such a drug or device during the course of this study
9. Pregnant females
10. Subject is unable to understand verbal and/or written English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2018-01-04 (Actual); Primary Completion 2019-10-10 (Actual); Study Completion 2020-10-10 (Actual)

PRIMARY OUTCOMES:
Knee Joint Chemical Profile | 1 week
  Evaluation of ELISA assay on synovial fluid aspirated pre and post study injection to ascertain the chemical profile of the joint for specific targets which include hyaluronic acid concentration, protein content and for increased levels of the following anabolic factors,IL1ra, TMP1, TMP2, HA, and IGF1 as well as decreased levels of the following degradative factors, IL-1, TNF-alpha, IL-10, MMP-2, MMP-9, TGF-beta5.

SECONDARY OUTCOMES:
VAS Pain scale | 1 week
  Measure self reported pain pre and post injection using Visual Analogue Scale rating 0 to 10, where 0 represents no pain and 10 represents worst imaginable pain.
Function | 1 week
  Measure self reported function pre and post injections using the validated Knee Injury and Osteoarthritis Outcome Score (KOOS).

CONTACTS AND LOCATIONS:
Overall Officials: Kevin R Stone, MD, Principal Investigator — The Foundation for Sports Medicine and Arthritis Research (Stone Research Foundation)
Locations (1):
- Stone Research Foundation, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No